CLINICAL TRIAL: NCT02596997
Title: An Intermediate-size, Expanded Access Protocol to Provide Brincidofovir for the Treatment of Serious Adenovirus Infection or Disease
Brief Title: Expanded Access Protocol to Provide Brincidofovir for the Treatment of Serious Adenovirus Infection or Disease
Status: No longer available | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CMX001-351
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2020-02

CONDITIONS: Adenovirus
Keywords: Adenovirus Brincidofovir
MeSH Terms: conditions — Adenoviridae Infections | interventions — brincidofovir

INTERVENTIONS:
Drug: Brincidofovir — Up to 100mg Brincidofovir twice weekly, not to exceed a total dose of 200mg each week
  Other Names: BCV CMX001

SUMMARY:
Provide patients with serious AdV infection or disease access to treatment with BCV.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed serious AdV infection based on clinical symptoms and laboratory testing showing AdV in the blood or other bodily fluids
* Able to swallow medication, either tablet or liquid

Exclusion Criteria:

* Previous dosing with Brincidofovir
* If female, not pregnant or trying to become pregnant

Min Age: 2 Months | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Children's Hospital LA, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Pediatric Stem Cell Transplantation Stanford University, Palo Alto, California
  - Stanford University, Palo Alto, California
  - UC San Diego Moores Cancer center, San Diego, California
  - University of California San Francisco Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - All Childrens Research Institute, St. Petersburg, Florida
  - All Children's Research Institute, St. Petersburg, Florida
  - Emory University-AFLAC Cancer and Blood Disorder Clinic, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Children's Mercy Hospital, Kansas City, Kansas
  - University of Louisville-Kosair Childrens Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Brigham & Woman's Hospital/Boston, Boston, Massachusetts
  - Michigan State/Spectrum Health, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Hackensack University MC, Hackensack, New Jersey
  - Weill Conrell Medical Center, New York, New York
  - Morgan Stanley Children's Hospital, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - New York Medical College-Maria Fareri Childrens hospital, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - New York Medical College, Maria Fareri Children's Hospital, Valhalla, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical System, Durham, North Carolina
  - Cincinnatti Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Childrens hospital of Philadelphia, Philadelphia, Pennsylvania
  - Methodist University Hospital-BMT program west clinic, Memphis, Tennessee
  - St. Jude Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Baylor College of Medicine-Infectious Disease, Houston, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Washington/ Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Wauwatosa, Wisconsin